CLINICAL TRIAL: NCT01094080
Title: Formula With Modified Content of Protein and Improved Fatty Acids and Their Impact on Infant Growth and Health
Acronym: BEMIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: HiPP GmbH & Co. Vertrieb KG (Industry)
Responsible Party: Principal Investigator, Prof. Berthold Koletzko, Prof, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 502042
Record Dates: First submitted 2010-02-01; First posted 2010-03-26 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Infant Nutrition
Keywords: fully formula fed; fully breast fed
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard infant formula (Active Comparator): infants are fed a commercial formula during the first 4 month of life, according to protocol
  Interventions: Other: standard infant formula
- modified infant formula (Experimental): infants are fed a modified infant formula (modified protein content and fatty acid pattern) during the first 4 month of life, according to protocol
  Interventions: Other: modified infant formula
- breast milk (Other): infants are breast fed
  Interventions: Other: breast milk

INTERVENTIONS:
Other: standard infant formula — infants are fed a commercial formula
  Arms: standard infant formula
Other: modified infant formula — the modified infant formula has a different protein content than the standard formula and long chain polyunsaturated fatty acids are added
  Arms: modified infant formula
Other: breast milk — infants are breast fed
  Arms: breast milk

SUMMARY:
In this study, the suitability of an infant formula with a modified content of protein and fatty acid pattern (LC-PUFA) for healthy term infants will be investigated.

Primary hypothesis to be tested is: an infant formula with a modified protein content is non inferior compared to a standard infant formula in respect to the growth of healthy term infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy term newborn
* gestational age between 37 and 41 weeks
* birth weight between the 3th and 97th weight-for-age percentile according to the EURO-Growth charts
* fully bottle-fed (at the latest with 28 days of age) or fully breast fed
* written parental informed consent
* Serbian nationality

Exclusion Criteria:

* malformations, congenital heart defect, congenital vascular disease, severe diseases of gastrointestinal tract, kidney, liver, central nervous system and/or metabolic disease
* intensive care during first 14 days of life
* participation in any other clinical study intervention
* twins, multiple birth
* neonatal infection
* medication and parenteral nutrition
* metabolic disorders
* birth-related complications
* severe disturbances of neonatal adaption

Ages: 3 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 505 (Actual)
Dates: Start 2010-02; Primary Completion 2011-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
change of weight from day 30 to day 120 | postnatal age 30 to 120 days

SECONDARY OUTCOMES:
anthropometry | postnatal day 30, day 60, day 90, day 120 days
  including body length, head circumference and derived parameter e.g. weight (from primary outcome) for length
blood markers | postnatal day 30, day 60, day 90, day 120 days (120 only)
Follow-up | 4 Years of age
  At 4 Years of Age, an Interview Regarding Severe Events and Growth Since Study End Will be Performed and Anthropometric Data (Weight, Length, Head Circumference and Body Composition Measured Via Skinfolds and BIA) Will be Collected.
Follow-up at age 7 years with an interview regarding severe events and growth | 7 years of age
  At 7 years of age we will perform anthropometric measurements (weight, height, head circumference and skinfolds) and bioimpedance measurement (from skinfolds and bioimpedance body composition will be estimated) additionally in an interview information on severe events (i.e. diseases) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Koletzko, Prof., Study Director — Hauner Children Hospital, Ludwig Maximilians Universität; Tatjana Nicolić Nicolić, Dr., Principal Investigator — Institute for Gynecology and Obstretition of Clinical Center Belgrade
Locations (2):
- Hauner Childrens Hospital, LudwigMaximilans Universität, München, Germany
- Institute for Gynecology and Obstretition of Clinical Center, Belgrade, Serbia

REFERENCES:
- [Result] Fleddermann M, Demmelmair H, Grote V, Nikolic T, Trisic B, Koletzko B. Infant formula composition affects energetic efficiency for growth: the BeMIM study, a randomized controlled trial. Clin Nutr. 2014 Aug;33(4):588-95. doi: 10.1016/j.clnu.2013.12.007. Epub 2013 Dec 30. PMID 24411489
- [Result] Fleddermann M, Demmelmair H, Grote V, Bidlingmaier M, Grimminger P, Bielohuby M, Koletzko B. Role of selected amino acids on plasma IGF-I concentration in infants. Eur J Nutr. 2017 Mar;56(2):613-620. doi: 10.1007/s00394-015-1105-9. Epub 2015 Nov 30. PMID 26621633